CLINICAL TRIAL: NCT07356531
Title: Clinical Trial Evaluating the Safety and Efficacy of Tumor Thermosensitive Embolic Agent in Transcatheter Arterial Chemoembolization for Primary Liver Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: JIANGSU SHENMING Medical Technology CO., Ltd (Industry)
Responsible Party: Sponsor
Organization: GrandPharma (China) Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SM-WMSSJ-001
Record Dates: First submitted 2025-11-26; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Liver Cancer
Keywords: thermosensitive embolic agent
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Intervention Model Description: This trial is a prospective, multicenter, randomized, parallel-controlled, non-inferiority clinical trial.
Masking Description: open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tumor thermosensitive embolic agent (Experimental): The experimental group received anthracycline chemotherapy drugs, iodinated oil, and tumor thermosensitive embolic agents。
  Interventions: Device: Transcatheter Arterial Chemoembolization
- Gelatin sponge granules embolic agent (Active Comparator): The control group received anthracycline chemotherapy drugs, iodinated oil, and gelatin sponge particle embolic agents
  Interventions: Device: Transcatheter Arterial Chemoembolization

INTERVENTIONS:
Device: Transcatheter Arterial Chemoembolization — In the main research stage, the researchers randomly confirmed the subject groups, and the experimental group used anthracycline chemotherapy drugs, iodized oil, and tumor thermosensitive embolization agents for embolization; The control group was treated with anthracycline chemotherapy drugs, iodized oil, and gelatin sponge particles embolization for embolization.
  Other Names: Tace

SUMMARY:
This is a prospective, multicenter, randomized, parallel-controlled, non-inferiority clinical trial that will be conducted at multiple clinical trial institutions in China. The trial is divided into two phases: the lead-in phase and the main study phase, with a total of 216 subjects planned to be enrolled. In the main study phase, subjects will be randomly assigned in a 1:1 ratio to either the test group or the control group. The randomly assigned subjects will receive TACE treatment. The test group will receive embolization therapy with anthracycline chemotherapy drugs, iodinated oil, and tumor temperature-sensitive embolic agents (test group), while the control group will receive embolization therapy with anthracycline chemotherapy drugs, iodinated oil, and gelatin sponge particles (control group).

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and effectiveness of the tumor thermosensitive he main efficacy evaluation indicator of this clinical trial is disease control rate. This indicator is widely regarded as a reflection of the effectiveness of tumor treatment, indicating the proportion of tumors that completely disappear, shrink, or remain stable after TACE treatment. Analyzing the results of the subjects, indirectly and directly reflecting clinical benefits, is preliminary reliable evidence of anti-tumor activity in treatment. As the main purpose of this experiment is to evaluate the tumor response of liver tumors treated with TACE using tumor thermosensitive embolic agents and compare it with gelatin sponge embolic agents,

ELIGIBILITY:
Inclusion Criteria:

* 1) Aged 18 to 80 (inclusive), of either gender;
* 2) Subjects who have been diagnosed with hepatocellular carcinoma (pathologically or clinically) according to the diagnostic criteria in the "Diagnosis and Treatment Guidelines for Primary Liver Cancer (2024 Edition)" and require TACE treatment;
* 3) Subjects with stage Ⅱb and Ⅲa liver cancer according to the Chinese Liver Cancer Staging Classification (CNLC), as well as subjects with stage Ⅰa, Ⅰb, and Ⅱa liver cancer who are not suitable/willing for surgical resection, liver transplantation, and ablation therapy;
* 4) Subjects with at least one untreated intrahepatic tumor lesion (maximum diameter ≤10cm) that meets the mRECIST definition (diameter ≥1cm);
* 5) The subjects agree to participate in this study and sign the informed consent form.

Exclusion Criteria:

* 1) Subjects whose target lesions have undergone local treatment (including but not limited to surgery, TACE, radiotherapy, hepatic artery infusion, ablation, etc.), or subjects whose target lesions require ablation/radiotherapy in combination with TACE treatment at the time of enrollment;
* 2) Subjects whose blood routine test results meet the following criteria: white blood cell count <3.0×10^9/L; platelet count <50×10^9/L, and this condition cannot be corrected (excluding subjects with hypersplenism or chemotherapy-induced bone marrow suppression);
* 3) Renal dysfunction: serum creatinine >176.8 μmol/L or creatinine clearance rate < 30 ml/min;
* 4) Uncorrectable coagulation dysfunction;
* 5) Uncorrectable hypercalcemia and respiratory acidosis;
* 6) Patients with systemic cachexia or multiple organ failure;
* 7) Patients with severe infections that cannot be effectively controlled and are not suitable for TACE treatment;
* 8) Complete obstruction of the main portal vein, insufficient collateral compensation of the portal vein, and inability to restore portal venous blood flow to the liver through portal veinoplasty;
* 9) Known contraindications or allergies to anthracycline chemotherapeutic drugs, calcium chloride injection, contrast media, and embolic materials;
* 10) Patients who are currently using cardiac glycosides;
* 11) Patients with target lesions who are at risk of ectopic embolism in the feeding artery (such as vascular access endangering normal areas, uncorrectable arteriovenous fistulas, and portal vein fistulas) or anatomical abnormalities that make them unsuitable for interventional procedures;
* 12) Patients who have been diagnosed with other malignant tumors within 2 years before randomization (except for basal cell or squamous cell skin cancer, cervical or breast carcinoma in situ that have been resected radically);
* 13) Patients with diffuse or distant extensive metastasis of tumors, with an expected survival time of less than 90 days;
* 14) Pregnant/lactating women, or those who have family planning;
* 15) Subjects who have participated in other drug or medical device intervention clinical trials within 30 days before randomization;
* 16) Other subjects who were considered unsuitable for participation in this clinical trial by the researchers.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2024-07-29 (Actual); Primary Completion 2025-11-14 (Actual); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
DCR | 30 days ± 7 days after the first TACE treatment
  Target lesion disease control rate

SECONDARY OUTCOMES:
Immediate success rate of target lesion embolization | Immediately after the initial TACE
  The immediate success rate of target lesion embolization refers to the percentage of successful embolization cases in the total number of cases immediately after the initial TACE angiography review.
Objective remission rate of target lesion | 30 days ± 7 days after the first TACE treatment, 30 days ± 7 days, 90 days ± 15 days and 180 days ± 30 days after the last TACE treatment
  Objective remission rate of target lesion
DCR | 30 days, 90 days and 180 days after the last TACE treatment
  Disease control rate of target lesions
Duration of target lesion response | 30 days after the first TACE treatment, 30 days, 90 days, and 180 days after the last TACE treatment
  The duration of target lesion response refers to the time from the initial recording to the target lesion CR or PR to the target lesion PD or death
AFP | 30 days ± 7 days after the first TACE treatment, 30 days ± 7 days, 90 days ± 15 days and 180 days ± 30 days after the last TACE treatment
  Changes of serum alpha fetoprotein values
Duration of embolization | Immediately after surgery
  the average value of the time taken for the embolization of a single lesion was calculated according to the number of embolic lesions
Embolization times | Within 90 days after surgery
  Record the total number of TACE treatments received by the subject from enrollment to the end of the trial
Device performance evaluation | within 1 day after surgery
  The surgeon conducted a subjective evaluation of the performance of the trial device during the surgical process after the operation, including system infusion performance, embolization performance, imaging performance, and overall evaluation, using a grading system of "excellent", "good", "fair", "acceptable", and "poor" to complete the evaluation

CONTACTS AND LOCATIONS:
Locations (15):
- China (15):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Affiliated Cancer Hospital of Guangxi Medical University, Nanning, Guangxi
  - The Affiliated Cancer Hospital of Guizhou Medical University, Guiyang, Guizhou
  - The Fourth Hospital of Hebei Medical University (Hebei Provincial Cancer Hospital), Shijiazhuang, Hebei
  - Anyang Tumor Hospital, Anyang, Henan
  - The First Affiliated Hospital of Henan University of Science & Technology, Luoyang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Yichang Central People's Hospital, Yichang, Hubei
  - First Affiliated Hospital of Gannan Medical University, Ganzhou, Jiangxi
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jilin Guowen Hospital, Gongzhuling, Jilin
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - Lishui Central Hospital, Lishui, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided